CLINICAL TRIAL: NCT05459701
Title: The Hepato-protective Effect of Dapagliflozin in Type 2 Diabetes Mellitus Patients (T2DM) With Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Dapagliflozin in Type 2 Diabetes Mellitus Patients (T2DM) With Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rehab Werida (Other)
Collaborators: University of Alexandria (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Associate Professor, Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dapagliflozin in NAFLD
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Nonalcoholic Fatty Liver Disease; Type 2 Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized (1:1), double-blind clinical trial, will be carried out on 50 patients who are candidate to detect the hepato-protective effect of Dapagliflozin on diabetic type 2 patients with non- alcoholic fatty disease (dapagliflozin 10 mg once daily for 24 - 48 weeks
  -Patients will be randomly allocated into two equal groups (25 patients each); group (A) for controlled (placebo), and the other group (D) for Dapagliflozin.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (A) for controlled (placebo). (Placebo Comparator): 25 patients will recieve placebo for 6 months.
  Interventions: Other: Placebo
- group (D) for Dapagliflozin. (Active Comparator): 25 patients will recieve 10 mg Dapagliflozin daily for 6 months.
  Interventions: Drug: Dapagliflozin 10mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10 mg once daily for 24 weeks.
  Other Names: Dapagliflozin 10 mg.
  Arms: group (D) for Dapagliflozin.
Other: Placebo — Placebo
  Arms: group (A) for controlled (placebo).

SUMMARY:
The aim of this study is to evaluate the effect of dapagliflozin on liver function of patient with NAFLD and T2DM.

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from Ethics committee of Faculty of Pharmacy, Damanhour University.
2. Ethical committee approval will be obtained from Ethics committee of General Organization for Teaching Hospitals and Institutes.
3. About 50 patients who are candidate to detect the hepato-protective effect of Dapagliflozin on non- alcoholic fatty disease, will be recruited from Alexandria Teaching Hospital (EL-Mery), General Organization for Teaching Hospitals and Institutes.
4. All participants should agree to take part in this clinical study and will provide informed consent.
5. Demographic data; age (year), sex (female/male), weight (kg), height (cm), BMI (kg/m2) will be collected.
6. Venous blood samples (5 ml will be collected by a sterile syringe then placed in a suitable sterile tube to be centrifuged, the serum will be reserved and stored at -80°C until the analysis) before, and after receiving medication (Dapagliflozin).
7. Measuring outcome:

   1. The biochemical tests will be done on the patients are alanine aminotransferase (ALT), aspartate aminotransferase (AST), homeostasis model assessment of insulin resistance (HOMA-IR), Hemoglobin A1C (HbA1C), Low-density lipoproteins (LDL), High-density lipoproteins (HDL), Triglycerides (TG), liver fibrosis score, and complete blood count (CBC).
   2. The molecular tests will be done on the patient are soluble vascular cell adhesion molecule-1 (Svcam-1), adipocytes (e.g. adiponectin, leptin).
8. The ultrasound screening will be done at first examination.
9. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
10. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus patients.
2. HbA1C < 8.5.
3. Patients were They were having fatty liver changes on abdominal ultrasound and mild to moderate elevation of serum liver enzymes.
4. BMI more than 30

Exclusion Criteria:

1. Patients with a history of alcohol, smoking, uncontrolled diabetes.
2. (HbA1c > 9.0).
3. Pregnancy.
4. Lactation.
5. Hemochromatosis.
6. Thyroid disorders.
7. Renal dysfunction.
8. Cardiac problem.
9. Chronic liver and decompensated liver disease in the form of hepatitis B and C.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
leptin (ng/ml) | 6 months
  leptin by enzyme-linked immunosorbent assay (ELISA).
adiponectin (pg/ml) | 6 months
  adiponectin by enzyme-linked immunosorbent assay (ELISA).
VCAM-1 (ng/ml) | 6 months
  VCAM-1 was analyzed in serum using the human VCAM-1 ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass Prof., Study Chair — Damanhour University; Amira B. Kassem, Lecturer, Principal Investigator — Damanhour University; Yasmin Essam, Bachlor, Principal Investigator — Damanhour University
Locations (1):
- Rehab Hussein Werida, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiba Y, Yamada T, Tsukita S, Takahashi K, Munakata Y, Shirai Y, Kodama S, Asai Y, Sugisawa T, Uno K, Sawada S, Imai J, Nakamura K, Katagiri H. Dapagliflozin, a Sodium-Glucose Co-Transporter 2 Inhibitor, Acutely Reduces Energy Expenditure in BAT via Neural Signals in Mice. PLoS One. 2016 Mar 10;11(3):e0150756. doi: 10.1371/journal.pone.0150756. eCollection 2016. PMID 26963613
- [Result] Tahara A, Kurosaki E, Yokono M, Yamajuku D, Kihara R, Hayashizaki Y, Takasu T, Imamura M, Li Q, Tomiyama H, Kobayashi Y, Noda A, Sasamata M, Shibasaki M. Effects of SGLT2 selective inhibitor ipragliflozin on hyperglycemia, hyperlipidemia, hepatic steatosis, oxidative stress, inflammation, and obesity in type 2 diabetic mice. Eur J Pharmacol. 2013 Sep 5;715(1-3):246-55. doi: 10.1016/j.ejphar.2013.05.014. Epub 2013 May 23. PMID 23707905
- [Result] Ohki T, Isogawa A, Toda N, Tagawa K. Effectiveness of Ipragliflozin, a Sodium-Glucose Co-transporter 2 Inhibitor, as a Second-line Treatment for Non-Alcoholic Fatty Liver Disease Patients with Type 2 Diabetes Mellitus Who Do Not Respond to Incretin-Based Therapies Including Glucagon-like Peptide-1 Analogs and Dipeptidyl Peptidase-4 Inhibitors. Clin Drug Investig. 2016 Apr;36(4):313-9. doi: 10.1007/s40261-016-0383-1. PMID 26914659